CLINICAL TRIAL: NCT02670083
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy And Safety Study of Crenezumab in Patients With Prodromal to Mild Alzheimer's Disease.
Brief Title: A Study Evaluating the Efficacy and Safety of Crenezumab Versus Placebo in Participants With Prodromal to Mild Alzheimer's Disease (AD).
Acronym: CREAD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was discontinued due to an interim analysis in this study, which indicated that Crenezumab was unlikely to meet its primary endpoint.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN29552; 2015-003034-27 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received intravenous (IV) infusion of Placebo every 4 weeks (Q4W) for 100 weeks.
  Interventions: Drug: Placebo
- Crenezumab (Experimental): Participants received intravenous (IV) infusion of Crenezumab every 4 weeks (Q4W) for 100 weeks.
  Interventions: Drug: Crenezumab

INTERVENTIONS:
Drug: Crenezumab — Crenezumab was administered by intravenous (IV) infusion at 60mg/kg as per the dosing schedule described above.
  Arms: Crenezumab
Drug: Placebo — Placebo was administered by intravenous (IV) infusion at 60mg/kg as per the dosing schedule described above.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group study will evaluate the efficacy and safety of crenezumab versus placebo in participants with prodromal to mild AD. Participants will be randomized 1:1 to receive either intravenous (IV) infusion of crenezumab or placebo every 4 weeks (Q4W) for 100 weeks. The final efficacy and safety assessment will be performed 52 weeks after the last crenezumab dose. Participants will then have the option to enter the Open Label Extension (OLE) study if eligible. Participants who do not enter the OLE study will have additional follow-up visits at 16 and 52 weeks after the last dose, primarily for safety and also for limited efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 40 and 120 kilograms (Kg) inclusive
* Availability of a person (referred to as the "caregiver") who in the investigator's judgment:
* Has frequent and sufficient contact with the participant to be able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits (which require partner input for scale completion), signs the necessary consent form, and has sufficient cognitive capacity to accurately report upon the participant's behavior and cognitive and functional abilities
* Fluency in the language of the tests used at the study site
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing (eye glasses and hearing aids are permitted)
* Evidence of the AD pathological process, by a positive amyloid assessment either on cerebrospinal fluid (CSF) amyloid beta 1-42 levels as measured on the Elecsys beta-amyloid(1-42) test system or amyloid PET scan by qualitative read by the core/central PET laboratory
* Demonstrated abnormal memory function at screening (up to 4 weeks before screening begins) or screening (FCSRT cueing index =<0.67 AND free recall =<27)
* Screening mini mental state examination (MMSE) score of greater than or equal to (>=) 22 points and Clinical Dementia Rating-Global Score (CDR-GS) of 0.5 or 1.0
* Meets National Institute on Aging/Alzheimer's Association (NIAAA) core clinical criteria for probable AD dementia or prodromal AD (consistent with the NIAAA diagnostic criteria and guidelines for mild cognitive impairment (MCI)
* If receiving symptomatic AD medications, the dosing regimen must have been stable for 3 months prior to screening
* Participant must have completed at least 6 years of formal education after the age of 5 years

Exclusion Criteria:

* Any evidence of a condition other than AD that may affect cognition such as other dementias, stroke, brain damage, autoimmune disorders (e.g. multiple sclerosis) or infections with neurological sequelae.
* History of major psychiatric illness such as schizophrenia or major depression (if not considered in remission)
* At risk of suicide in the opinion of the investigator
* Any abnormal MRI findings, such as presence of cerebral vascular pathology, cortical stroke, etc or inability to tolerate MRI procedures or contraindication to MRI
* Unstable or clinically significant cardiovascular (e.g., myocardial infarction), kidney or liver disease
* Uncontrolled hypertension
* Screening hemoglobin A1c (HbA1C) >8%
* Poor peripheral venous access
* History of cancer except:

If considered to be cured or If not being actively treated with anti-cancer therapy or radiotherapy

- Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (196):
- United States (66):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Pharmacology Research Inst, Encino, California
  - Collaborative Neuroscience Network Inc., Long Beach, California
  - Alliance for Wellness, dba Alliance for Research, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - USC Keck School Of Medicine, Los Angeles, California
  - UCLA Medical Center, Department of Neurology, Los Angeles, California
  - Pharmacology Research Inst, Newport Beach, California
  - Shankle Clinic, Newport Beach, California
  - Stanford Univ Medical Center, Palo Alto, California
  - Anderson Clinical Research, Inc., Redlands, California
  - University of California, Davis; Alzheimers Disease Center, Department of Neurology, Sacramento, California
  - UCSF - Memory and Aging Center, San Francisco, California
  - Neurological Research Inst, Santa Monica, California
  - North Bay Neuro Science Institute, Sebastopol, California
  - Associated Neurologists PC - Danbury, Danbury, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Bradenton Research Center, Bradenton, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Galiz Research, LLC, Hialeah, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Merritt - Island Medical Research, Merritt Island, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Bioclinica Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Johnnie B. Byrd Sr. Alzheimer's Center & Research Institute, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Compass Research, The Villages, Florida
  - Emory University, Atlanta, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - MidAmerica Neuroscience Institute, Prairie Village, Kansas
  - Maine Research Associates, Auburn, Maine
  - MMP Neurology, Scarborough, Maine
  - Springfield Neurology Associates, Springfield, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Albany Medical Faculty Physicians COmmunity Division. The Neurology Group, Albany, New York
  - Neurological Associates of Albany, PC, Albany, New York
  - Dent Neurological Institute, Amherst, New York
  - Columbia University Medical Center, New York, New York
  - South Shore Neurologic Associates P.C., Patchogue, New York
  - Behavioral Health Research, Charlotte, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Insight Clinical Trials LLC, Shaker Heights, Ohio
  - Oklahoma Clinical Research, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Central States Research, Tulsa, Oklahoma
  - Summit Research Network Inc., Portland, Oregon
  - Drexel Univ College of Med; Clinical Research Group, Philadelphia, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Senior Adults Specialty Research, Austin, Texas
  - Kerwin Research Center, LLC, Dallas, Texas
  - University of North Texas Health Science Center; Fort Worth Patient Care Center, Fort Worth, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
  - Caulfield Hospital; Aged Psychiatry Research Unit, Caulfield, Victoria
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Neurodegenerative Disorders Research; Neurology, West Perth, Western Australia
- Konventhospital Barmherzige Brüder; Neurologie I, Linz, Austria
- UZ Gent, Ghent, Belgium
- Bulgaria (2):
  - ACIBADEM CITY CLINIC TOKUDA HOSPITAL EAD; Clinic of Neurology and Sleep Medicine, Sofia
  - Alexandrovska hospital; Neurology Department, Sofia
- Canada (9):
  - Vancouver Hospital - UBC Hospital Site, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Parkwood Hospital; Geriatric Medicine, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - CHA Hopital de I enfant-Jesus, Québec, Quebec
- Costa Rica (2):
  - Hospital Clínica Biblica, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- Clinical Hospital Centre Zagreb;Clinic for Neurology, Zagreb, Croatia
- Czechia (2):
  - Charles University, Medical faculty, Hradec Kralove ;Department of Neurology, Hradec Králové
  - General Teaching Hospital, Departmetn of Neurology, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Neurologisk Afdeling F, Demensklinikken, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
- Finland (2):
  - Terveystalo Tampere, Tampere
  - CRST Oy, Turku
- France (7):
  - Hopital Avicenne; Neurologie, Bobigny
  - Hopital neurologique Pierre Wertheimer - CHU Lyon; Neurologie, Bron
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - Hopital Lariboisiere, Paris
  - CHU Poitiers - Hopital La Miletrie, Poitiers
  - Hopital Hautepierre; Centre dInvestigation Clinique, Strasbourg
  - CHU Toulouse - La Grave, Toulouse
- Germany (8):
  - Neurologische Praxis Dr. Andrej Pauls, München
  - Klinikum rechts der Isar der TU München; Klinik für Psychiatrie und Psychotherapie, München
  - Universitätsklinikum Münster; Klinik und Poliklinik für Neurologie, Münster
  - Steinwachs Klaus; Arztpraxis fur Neurologie u. Psychiatrie, Nuremberg
  - Universitätsklinikum Rostock Zentrum für Nervenheilkunde, Rostock
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
  - Studienzentrum Nordwest, Dr. med. Joachim Springub / Herr Wolfgang Schwarz, Westerstede
  - Forschungszentrum Ruhr, Witten
- Hong Kong (2):
  - Prince of Wales Hospital; Dept. of Medicine & Therapeutics, Hong Kong
  - Queen Mary Hospital, Division of Geriatric Medicine, Hong Kong
- Hungary (5):
  - Semmelweis University; Department of Neurology, Budapest
  - Szabolcs-Szatmár-Bereg Megyei Kórházak - Jósa András Oktatókórház; Pszichiátria, Nyíregyháza
  - University of Szeged; Department of Psychiatry, Szeged
  - Szent Borbala Korhaz; Neurologiai es Stroke Osztaly, Tatabánya
  - Jávorszky Ödön Kórház, Neurológia és stroke osztály, Vác
- Italy (7):
  - Fondazione Santa Lucia IRCCS; Neurologia e Riabilitazione Neurologica, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratell;Neurologia, Rome, Lazio
  - Ente Ospedaliero Ospedali Galliera; Ambulatorio di Neurologia, Genoa, Liguria
  - Casa di Cura Policlinico; Dipartimento di Scienze Neuroriabilitative, Milan, Lombardy
  - Ospedale S. Maria Nascente; Fondazione Don Gnocchi; Dip. Neurologia Riabilitativa, Milan, Lombardy
  - Ospedale Casati Passirana di Rho; Centro Regionale Alzheimer, Passirana, Lombardy
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; S.C. Geriatria, Perugia, Umbria
- Japan (10):
  - Miyoshi Clinic of Neurology, Hananosato, Hiroshima
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Rakuwakai Otowarehabilitation Hospital, Kyoto
  - Mie University Hospital, Mie
  - National Hospital Organization Matsumoto Medical Center, Nagano
  - Saigata Medical Center, Niigata
  - Katayama Medical Clinic, Okayama
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
- Vilnius University Hospital Santariskiu Clinic, Vilnius, Lithuania
- Mexico (4):
  - Hospital Angeles de Culiacán, Neurociencias Estudios Clínicos SC, Culiacán
  - Hospital Uni; Dr. Jose E. Gonzalez, Monterrey
  - AVIX Investigación Clínica S.C, Monterrey
  - Hospital Universitario de Saltillo, Saltillo
- Poland (6):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - NZOZ NEURO-KARD Ilkowski i Partnerzy Sp. Partn. Lek, Poznan
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - Przychodnia Specjalistyczna PROSEN, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - Optimum, Warsaw
- Portugal (2):
  - Hospital Prof. Dr. Fernando Fonseca; Servico de Neurologia, Amadora
  - Hospital Beatriz Angelo; Servico de Neurologia, Loures
- Russia (7):
  - State Autonomous Healthcare Institution "Republican Clinical Neurological Center, Kazan'
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan'
  - Institution of RAMS (Mental Health Research Center of RAMS), Moscow
  - SBEI of HPI The 1st Moscow State Medical University n.a. I.M. Sechenov of MOH of RF, Moscow
  - SHI City Psychoneurological Dispensary #7, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M.Kirov; Neurology Department, Saint Petersburg
  - City Clinical Hospital # 2 n.a. V.I. Razumovsky, Saratov
- University Medical Centre Maribor, Maribor, Slovenia
- South Korea (6):
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - KyungHee Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital; Dept of Neurology, Seoul
- Spain (19):
  - Fundació ACE, BArcelon, Barcelona
  - Hospital Universitari de Bellvitge; Servicio de Neurologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Sant Joan de Deu; Servicio de Neurología, Manresa, Barcelona
  - Hospital General De Catalunya; Servicio de Neurologia, Sant Cugat del Vallès, Barcelona
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital Virgen del Puerto. Servicio de Neurología, Plasencia, Caceres
  - Hospital Universitario Marques de Valdecilla; Servicio de Neurología, Santander, Cantabria
  - Clinica Universitaria de Navarra; Servicio de Neurología, Pamplona, Navarre
  - Complejo Asistencial Universitario de Salamanca; Servicio de Psiquiatría, Salamaca, Salamanca
  - Hospital General Universitario de Albacete; Servicio de Neurología, Albacete
  - Hospital Vall d'Hebron; Servicio de Neurología, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Clinica Ruber, 4 planta; Servicio de Neurologia, Madrid
  - Universitario de La Princesa; Servicio de Neurología, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Neurologia, Málaga
  - Hospital Universitario Virgen de Arrixaca; Servicio de Neurología, Murcia
  - Hospital Universitario la Fe; Servicio de Neurologia, Valencia
  - Servicio de Neurología Hospital Viamed Montecanal., Zaragoza
- Sweden (3):
  - Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo
  - Sahlgrenska Academy University,Neuroscience and Physiology;Departmt of Psychiatry and Neurochemistry, Mölndal
  - Karolinska Uni Hospital, Huddinge; Dept. of Geriatric Med, Stockholm
- Universitäres Zentrum für Altersmedizin und Rehabilitation, Basel, Switzerland
- Turkey (Türkiye) (4):
  - Hacettepe University School of Medicine; Neurology, Ankara
  - Osmangazi University School of Medicine,Neurology Department, Eskişehir
  - Istanbul University Istanbul School of Medicine; Neurology, Istanbul
  - Ondokuz Mayis University School of Medicine; Neurology, Samsun
- Ukraine (3):
  - Regional mental hospital; Department of psychiatry, psychology and sexology, Lviv, KIEV Governorate
  - National Medical Academy of Postgraduate Education named after P.L.Shupik; Neurology Department #1, Kiev
  - D.F.Chebotarev Institute of Gerontology NAMS;Depart of Age Physiology&Pathology of Nervous System, Kiev
- United Kingdom (8):
  - Royal Preston Hospital, Blackburn
  - Surrey and Borders NHS Foundation Trust; Brain Science Research Unit, Chertsey
  - Coventry and Warwickshire Partnership NHS Trust, Coventry
  - St George's Hospital, London
  - Charing Cross Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Campus for Ageing and Vitality, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Hibar DP, Bauer A, Rabe C, Borlinghaus N, Jethwa A, Kollmorgen G, Di Domenico A, Zetterberg H, Blennow K, Masters CL, Sperling RA, Bittner T. Elecsys pTau217 plasma immunoassay detection of amyloid pathology in clinical cohorts. Alzheimers Dement. 2026 Jan;22(1):e71009. doi: 10.1002/alz.71009. PMID 41537338
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Teng E, Manser PT, Shah M, Pickthorn K, Hu N, Djakovic S, Swendsen H, Blendstrup M, Faccin G, Ostrowitzki S, Sink KM. The Use of Episodic Memory Tests for Screening in Clinical Trials for Early Alzheimer's Disease: A Comparison of the Free and Cued Selective Reminding Test (FCSRT) and the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). J Prev Alzheimers Dis. 2023;10(1):41-49. doi: 10.14283/jpad.2022.101. PMID 36641609
- [Derived] Ostrowitzki S, Bittner T, Sink KM, Mackey H, Rabe C, Honig LS, Cassetta E, Woodward M, Boada M, van Dyck CH, Grimmer T, Selkoe DJ, Schneider A, Blondeau K, Hu N, Quartino A, Clayton D, Dolton M, Dang Y, Ostaszewski B, Sanabria-Bohorquez SM, Rabbia M, Toth B, Eichenlaub U, Smith J, Honigberg LA, Doody RS. Evaluating the Safety and Efficacy of Crenezumab vs Placebo in Adults With Early Alzheimer Disease: Two Phase 3 Randomized Placebo-Controlled Trials. JAMA Neurol. 2022 Nov 1;79(11):1113-1121. doi: 10.1001/jamaneurol.2022.2909. PMID 36121669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 249 centers in 30 countries.
Pre-assignment Details: A total of 813 participants were enrolled at 249 centers. 4 participants did not receive any study treatment meaning that the modified intent-to-treat and safety populations both consisted of 809 participants.
Period: Overall Study
Arm/Group | Placebo | Crenezumab
Started | 409 | 404
Completed | 88 | 85
Not Completed | 321 | 319
Not completed — Adverse Event | 16 | 13
Not completed — Death | 4 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Multiple Reasons | 9 | 9
Not completed — Physician Decision | 0 | 2
Not completed — Study Terminated By Sponsor | 257 | 254
Not completed — Symptomatic Deterioration | 0 | 2
Not completed — Withdrawal by Subject | 32 | 31
Not completed — Non-Compliance With Study Drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Crenezumab | Total
Number analyzed (Participants) | 409 | 404 | 813
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (8.4) | 71.0 (7.9) | 70.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 236 | 483
  Male | 162 | 168 | 330
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 39 | 32 | 71
  Not Hispanic or Latino | 361 | 369 | 730
  Not Stated | 7 | 2 | 9
  Unknown | 2 | 1 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 5 | 10 | 15
  Asian | 28 | 28 | 56
  Black or African American | 3 | 5 | 8
  Multiple | 0 | 1 | 1
  Unknown | 13 | 8 | 21
  White | 360 | 352 | 712

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 105 in Clinical Dementia Rating-Sum of Boxes (CDR-SB) Score
Description: The CDR-SB rates impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment = 0, questionable impairment = 0.5 and mild, moderate and severe impairment = 1, 2 and 3 respectively. The score range is from 0 to 18 with a high score indicating a high disease severity. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline for this primary endpoint. Data after 29 January 2019 are censored for the primary and secondary efficacy analyses to avoid potential biases due to investigators, participants, raters, etc. being potentially influenced by early closure of the study due to lack of efficacy.
Time Frame: Baseline, Week 105
Population: The Modified Intent-To-Treat population (Placebo (n = 407); Cren (n = 402)) was defined as all randomized participants who received at least 1 dose of study drug, with participants grouped according to the treatment assigned at randomization. Data presented below is only for participants that were included in the actual analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 88 | 86
Units on a Scale | 3.42 (0.263) | 3.59 (0.264)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.86 to 0.53], Standard Error of Mean 0.354

2. Secondary Outcome: Change From Baseline to Week 105 on Cognition, as Assessed by Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog) (Subscale) 13 (ADAS-Cog-13)
Description: The ADAS-Cog-13 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Most of these are assessed by tests although some are rated by the clinician on a 5-point scale. The ADAS-Cog-13 is the ADAS-Cog-11 with 2 further items: delayed word recall and total digit cancellation. The score range for ADAS-Cog-13 is from 0 to 85 with high scores representing severe dysfunction. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 86 | 80
Units on a Scale | 9.55 (0.824) | 9.82 (0.841)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.26, 95% CI 2-sided [-2.39 to 1.87], Standard Error of Mean 1.083

3. Secondary Outcome: Change From Baseline to Week 105 on Cognition, as Assessed by Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog) (Subscale) 11 (ADAS-Cog-11)
Description: The ADAS-Cog-11 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Most of these are assessed by tests although some are rated by the clinician on a 5-point scale. The score range for ADAS-Cog-11 is from 0 to 70 with high scores representing severe dysfunction. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 86 | 80
Units on a Scale | 8.43 (0.758) | 8.53 (0.773)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-2.08 to 1.88], Standard Error of Mean 1.006

4. Secondary Outcome: Change From Baseline to Week 105 on Severity of Dementia, Assessed Using the CDR-Global Score (CDR-GS)
Description: The CDR-GS represents a semi-structured interview which rates impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care) on a 5-point scale in which CDR 0 = no dementia and CDR 0.5, 1, 2 or 3 = questionable, mild, moderate or severe dementia respectively. The range in scores for the CDR-GS is from 0 to 3 and a high score on the CDR-GS would indicate a high disease severity. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 88 | 86
Units on a Scale | 0.55 (0.056) | 0.50 (0.056)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.05, 95% CI 2-sided [-0.10 to 0.20], Standard Error of Mean 0.076

5. Secondary Outcome: Change From Baseline to Week 105 on Severity of Dementia, Assessed Using the Mini Mental State Evaluation (MMSE)
Description: The MMSE is a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target 6 areas: orientation, registration, attention, short-term recall, language and constructional praxis/visuospatial abilities. The scores on the MMSE range from 0 to 30, with higher scores indicating better function. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 90 | 87
Units on a Scale | -4.63 (0.377) | -4.96 (0.383)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.33, 95% CI 2-sided [-0.62 to 1.29], Standard Error of Mean 0.486

6. Secondary Outcome: Change From Baseline to Week 105 on Function as Assessed by the ADCS-ADL Total Score
Description: The ADCS-ADL (Alzheimer's Disease Cooperative Study-Activities of Daily Living) is the scale most widely used to assess functional outcomes in participants with AD. The ADCS-ADL covers both basic ADL (e.g., eating and toileting) and more complex 'instrumental' ADL or iADL (e.g., using the telephone, managing finances and preparing a meal). The ADCS-ADL consists of 23 questions with a score range of 0 to 78 where a higher score represents better function. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 90 | 88
Units on a Scale | -11.51 (1.226) | -13.39 (1.242)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 1.88, 95% CI 2-sided [-1.43 to 5.18], Standard Error of Mean 1.679

7. Secondary Outcome: Change From Baseline to Week 105 on Function as Assessed by the ADCS-instrumental (ADCS-iADL) Subscore
Description: The ADCS-iADL (Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living) measures activities such as using the telephone, managing finances and preparing a meal. The ADCS-iADL consists of 16 questions with a score range of 0 to 56 where a higher score represents better function. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 90 | 88
Units on a Scale | -9.22 (0.967) | -10.44 (0.979)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 1.22, 95% CI 2-sided [-1.35 to 3.79], Standard Error of Mean 1.306

8. Secondary Outcome: Change From Baseline to Week 105 on a Measure of Dependence Derived From the ADCS-ADL Score
Description: as for outcome 6
Time Frame: Baseline, Week 105
Population: Please note that for this Outcome Measure, no participants were evaluated at all as the derivation of this endpoint was not pre-specified before the Sponsor terminated the study and therefore it was not reported.
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline to Week 105 Assessed Using the Neuropsychiatric Inventory Questionnaire (NPI-Q)
Description: The NPI-Q is an informant-based instrument that evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavioral disturbances and appetite and eating abnormalities. The severity of each neuropsychiatric symptom is rated on a 3-point scale (mild, moderate and marked). The total severity score range is from 0 to 36 with higher scores representing higher severity. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 84 | 87
Units on a Scale | 1.02 (0.562) | 1.55 (0.556)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.53, 95% CI 2-sided [-1.95 to 0.90], Standard Error of Mean 0.723

10. Secondary Outcome: Quality of Life-Alzheimer's Disease (QoL-AD) Scale Score
Description: The QoL-AD (Quality of Life - Alzheimer's Disease) scale assesses QoL in participants who have dementia. The QoL-AD consists of 13 items covering aspects of participants' relationships with friends and family, physical condition, mood, concerns about finances and overall assessment of QoL. Items are rated on 4-point Likert-type scales ranging from 1 [poor] to 4 [excellent]. The score range is from 13 to 52, with higher scores indicating a better QoL. The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline up to Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 90 | 86
Units on a Scale | -1.69 (0.501) | -2.08 (0.513)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.40, 95% CI 2-sided [-0.81 to 1.60], Standard Error of Mean 0.609

11. Secondary Outcome: Zarit Caregiver Interview for Alzheimer's Disease (ZCI-AD) Scale Score
Description: The ZCI-AD is a modified version of the Zarit Burden Interview, which was originally designed to reflect the stresses experienced by caregivers of people with dementia. This modified version includes slight modifications in item and title wording (e.g., removal of "your relative" to refer directly to the patient, removal of "burden" from title) and the use of 11-point numerical rating scales. The ZCI-AD scale consists of a total of 30 items. Total scores will be calculated with a total score range from 0 to 300 (higher scores indicate a higher burden on the caregiver). The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline up to Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 86 | 87
Units on a Scale | 22.72 (5.135) | 24.11 (5.106)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -1.39, 95% CI 2-sided [-13.64 to 10.86], Standard Error of Mean 6.214

12. Secondary Outcome: EQ-5D Questionnaire Domain Score for Participants
Description: The EQ-5D is a standardized measure of health status designed to provide a simple generic measure of health for clinical and economic appraisal. It is broadly applicable across a wide range of health conditions and treatment. The EQ-5D assesses five domains to provide a health state index. These are anxiety/depression, pain/discomfort, usual activities, mobility, and self-care. The scores on the EQ-5D ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). The difference in mean change from Baseline to Week 105 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline up to Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 89 | 87
Units on a Scale | -4.54 (1.732) | -6.35 (1.761)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 1.82, 95% CI 2-sided [-2.64 to 6.27], Standard Error of Mean 2.260

13. Secondary Outcome: EQ-5D Questionnaire Domain Score for Caregivers
Description: as for outcome 12
Time Frame: Baseline up to Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 89 | 88
Units on a Scale | -3.16 (1.713) | -4.09 (1.721)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.94, 95% CI 2-sided [-3.45 to 5.32], Standard Error of Mean 2.222

14. Secondary Outcome: Percentage of Participants With Adverse Event (AEs) and Serious Adverse Event (SAEs)
Description: An Adverse Event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up until 16 weeks after the last dose of study drug (up to 117 weeks).
Population: The Safety analysis population included all randomized participants who received at least 1 dose of study drug with participants grouped according to actual treatment received. If a participant received at least 2 vials of crenezumab, then they were placed in the crenezumab arm.
Measure: Number; unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 405 | 404
Percentage
  AEs | 83.2 | 85.9
  SAEs | 15.6 | 16.6

15. Secondary Outcome: Percentage of Participants With Anti-Crenezumab Antibodies
Description: Participants were considered positive or negative for ADA based on their baseline and post-baseline sample results. The number and percentage of participants with confirmed positive ADA levels were determined for Crenezumab and Placebo groups. The prevalence of ADA at baseline was calculated as the proportion of participants with confirmed positive ADA levels at baseline relative to the total number of participants with a sample available at baseline. The incidence of treatment-emergent ADAs was determined as the proportion of participants with confirmed post-baseline positive ADAs relative to the total number of participants that had at least one post-baseline sample available for ADA analysis.
Time Frame: Baseline up to Week 105
Population: The Safety analysis population included all randomized participants who received at least 1 dose of study drug with participants grouped according to actual treatment received. If a participant received at least 2 vials of crenezumab, then they were placed in the crenezumab arm. Data below is only for participants included in the actual analysis.
Measure: Number; unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 385 | 404
Percentage
  Baseline ADAs | 0.3 | 0.2
  Treatment Emergent ADAs: number analyzed (Participants) | 382 | 397
  Treatment Emergent ADAs | 0.5 | 0.5

16. Secondary Outcome: Serum Concentration of Crenezumab
Description: Serum concentration data for Crenezumab will be tabulated and summarized. Descriptive summary statistics will include the arithmetic mean and SD. Since a sparse PK sampling design is being used, population (non-linear mixed-effects) modeling will be used to analyze the dose concentration-time data of crenezumab. Information from other clinical studies may be incorporated to establish the PK model. Please note that Post-dose samples were not collected at Weeks 37 and 105.
Time Frame: Pre-infusion (0 hour), 60-90 minutes post-infusion on Day 1 Week 1 and on Week 25; Weeks 13, 37 (Pre-dose), 53, 77 and 105 (infusion length = as per the Pharmacy Manual)
Population: The PK Analysis population was defined as all participants who have received at least one dose of crenezumab and with at least one evaluable post-dose PK sample. Data presented below is only for participants that were included in the actual analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Crenezumab
Number analyzed (Participants) | 392
ug/mL
  Week 1 Day 1 Predose | NA (NA) — No Drug was administered at this point so no concentrations detected.
  Week 1 Day 1 Postdose: number analyzed (Participants) | 74
  Week 1 Day 1 Postdose | 1350 (319)
  Week 13 Predose: number analyzed (Participants) | 388
  Week 13 Predose | 345 (146)
  Week 13 Postdose: number analyzed (Participants) | 384
  Week 13 Postdose | 1580 (487)
  Week 25 Predose: number analyzed (Participants) | 378
  Week 25 Predose | 369 (130)
  Week 25 Postdose: number analyzed (Participants) | 54
  Week 25 Postdose | 1700 (443)
  Week 37 Predose: number analyzed (Participants) | 366
  Week 37 Predose | 368 (152)
  Week 53 Predose: number analyzed (Participants) | 363
  Week 53 Predose | 393 (164)
  Week 53 Postdose: number analyzed (Participants) | 60
  Week 53 Postdose | 1800 (420)
  Week 77 Predose: number analyzed (Participants) | 263
  Week 77 Predose | 410 (261)
  Week 77 Postdose: number analyzed (Participants) | 50
  Week 77 Postdose | 1790 (496)
  Week 105: number analyzed (Participants) | 89
  Week 105 | 408 (186)

17. Secondary Outcome: Plasma Amyloid Beta (Abeta) 40 Concentrations
Description: Plasma Abeta 40 concentrations will be measured over time and descriptive summary statistics will include the arithmetic mean and SD. Please note that a Post-dose sample was only collected at Week 13.
Time Frame: Week 1 Day 1; Weeks 13, 25, 53, 77 and 105
Population: The PD Analysis population was defined as all participants who have received at least one dose of crenezumab and with at least one evaluable post-dose PK sample. Data presented below is only for participants that were included in the actual analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crenezumab
Number analyzed (Participants) | 101
ng/mL
  Week 1 Day 1 Predose | 0.377 (0.136)
  Week 13 Predose: number analyzed (Participants) | 20
  Week 13 Predose | 44.6 (10.0)
  Week 13 Postdose: number analyzed (Participants) | 21
  Week 13 Postdose | 44.3 (9.5)
  Week 25 Predose: number analyzed (Participants) | 46
  Week 25 Predose | 46.4 (10.1)
  Week 53 Predose: number analyzed (Participants) | 94
  Week 53 Predose | 48.8 (10.7)
  Week 77 Predose: number analyzed (Participants) | 40
  Week 77 Predose | 47.5 (12.2)
  Week 105 Predose: number analyzed (Participants) | 38
  Week 105 Predose | 48.6 (14.0)

18. Secondary Outcome: Plasma Amyloid Beta (Abeta) 42 Concentrations
Description: Plasma Abeta 42 concentrations will be measured over time and descriptive summary statistics will include the arithmetic mean and SD. Please note that a Post-dose sample was only collected at Week 13.
Time Frame: Week 1 Day 1; Weeks 13, 25, 53, 77 and 105
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crenezumab
Number analyzed (Participants) | 101
ng/mL
  Week 1 Day 1 Predose | 0.0335 (0.00812)
  Week 13 Predose: number analyzed (Participants) | 20
  Week 13 Predose | 2.72 (0.553)
  Week 13 Postdose: number analyzed (Participants) | 21
  Week 13 Postdose | 2.71 (0.602)
  Week 25 Predose: number analyzed (Participants) | 46
  Week 25 Predose | 2.73 (0.55)
  Week 53 Predose: number analyzed (Participants) | 94
  Week 53 Predose | 2.87 (0.589)
  Week 77 Predose: number analyzed (Participants) | 40
  Week 77 Predose | 2.79 (0.68)
  Week 105 Predose: number analyzed (Participants) | 38
  Week 105 Predose | 2.87 (0.818)

19. Secondary Outcome: Percentage Change From Baseline to Week 105 in Whole Brain Volume as Determined by Magnetic Resonance Imaging (MRI)
Description: Percentage Change in Whole Brain Volume will be measured over time and descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 180 | 172
Percentage | -2.66 (0.091) | -2.65 (0.092)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.24 to 0.22], Standard Error of Mean 0.116

20. Secondary Outcome: Percentage Change From Baseline to Week 105 in Ventricle Volume as Determined by Magnetic Resonance Imaging (MRI)
Description: Percentage Change in Ventricle Volume will be measured over time and descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 189 | 181
Percentage | 22.29 (0.907) | 23.57 (0.912)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -1.28, 95% CI 2-sided [-3.72 to 1.17], Standard Error of Mean 1.245

21. Secondary Outcome: Percentage Change From Baseline to Week 105 in Hippocampal Volume as Determined by Magnetic Resonance Imaging (MRI)
Description: Percentage Change in Hippocampal Volume will be measured over time and descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 169 | 160
Percentage | -6.57 (0.200) | -6.97 (0.203)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.39, 95% CI 2-sided [-0.10 to 0.89], Standard Error of Mean 0.253

ADVERSE EVENTS:
Time Frame: Baseline up until 16 weeks after the last dose of study drug (up to 117 weeks).
Arm/Group | Placebo | Crenezumab
All-Cause Mortality (participants affected / at risk) | 5/405 | 8/404
Serious Adverse Events (participants affected / at risk) | 63/405 | 67/404
Other Adverse Events (participants affected / at risk) | 214/405 | 225/404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=405) | Crenezumab (N=404)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 2 (2) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM PRIMARY (Endocrine disorders) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (3)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL VASCULAR MALFORMATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
CHEST PAIN (General disorders) | 0 (0) | 2 (3)
DEATH (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 3 (3) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3) | 5 (5)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 2 (2)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
TUBERCULOSIS OF CENTRAL NERVOUS SYSTEM (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 3 (4) | 4 (5)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
SYSTEMIC SCLERODERMA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 2 (2)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 2 (3) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 2 (2)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 4 (4) | 3 (3)
DEVICE FAILURE (Product Issues) | 0 (0) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 2 (2)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DELUSION (Psychiatric disorders) | 0 (0) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 1 (1)
PERSONALITY CHANGE (Psychiatric disorders) | 0 (0) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (3)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE INTERSTITIAL PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 (1) | 0 (0)
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 1 (1) | 0 (0)
URETHRAL STENT INSERTION (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=405) | Crenezumab (N=404)
DIARRHOEA (Gastrointestinal disorders) | 26 (42) | 25 (27)
BRONCHITIS (Infections and infestations) | 13 (13) | 21 (21)
NASOPHARYNGITIS (Infections and infestations) | 33 (41) | 40 (50)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 29 (38) | 33 (36)
URINARY TRACT INFECTION (Infections and infestations) | 22 (29) | 20 (22)
FALL (Injury, poisoning and procedural complications) | 33 (42) | 42 (60)
WEIGHT DECREASED (Investigations) | 11 (11) | 22 (22)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 31 (36) | 26 (38)
DIZZINESS (Nervous system disorders) | 27 (34) | 23 (28)
HEADACHE (Nervous system disorders) | 45 (60) | 39 (48)
ANXIETY (Psychiatric disorders) | 21 (24) | 28 (31)
DEPRESSION (Psychiatric disorders) | 27 (27) | 28 (28)
RASH (Skin and subcutaneous tissue disorders) | 22 (26) | 7 (8)
HYPERTENSION (Vascular disorders) | 22 (22) | 27 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT02670083/Prot_SAP_000.pdf